CLINICAL TRIAL: NCT04008641
Title: Pertinence of Pediatric Message Delivered to Parents During Antenatal Consultations
Acronym: INFONEO
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Jean-Michel HASCOET, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: PSS2018/INFONEO-HASCOET/NK
Record Dates: First submitted 2019-06-04; First posted 2019-07-05 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Information Understanding and Psychological Impact
Keywords: pediatric consultation; psychological; comprehension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parents after pediatric antenatal consultation: Survey after pediatric antenatal consultation, for both members of couple if possible
  Interventions: Other: Pediatric consultation's survey

INTERVENTIONS:
Other: Pediatric consultation's survey — Realization of a pediatric consultation. At the end, evaluation of comprehension and psychological impact with a survey (completed by parents).

SUMMARY:
Antenatal consultations are experienced as traumatic for many couples. Moreover, when informations are given urgently ; comprehension and psychological impact aren't well evaluate.

This project aims to evaluate comprehension and psychological impact, for both members of the couple, when informations are provided urgently or during usual consultations.

ELIGIBILITY:
Inclusion Criteria:

* Parents whom pregnancies need antenatal pediatric consultation
* Non opposition

Exclusion Criteria:

* < 18 years old
* Psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All parents with need antenatal pediatric urgently or usual consultation
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Comprehension and psychological impact ; urgently informations compared with usual consultations | At pregnancy follow-up visit up to 36 weeks gestation
  After non opposition, surveys are given to parents
  Scale built by investigators. With items about comprehension and psychological impact. From 0 to 23. One point per item. Higher values (23/23) represent a better outcome (comprehension and good psychological impact (0/23 if not)).

SECONDARY OUTCOMES:
Difference between both members of the couple | At pregnancy follow-up visit up to 36 weeks gestation
  Same survey for both members, evaluation and comparison of answers.
  Same scale
Comprehension and psychological impact, at pregnancy's theoric term compared with first survey Same scale | At delivery at 41 weeks gestation
  Same survey, realized at pregnancies' theoric terms

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel HASCOET, MD, PhD, Principal Investigator — CHRU NANCY - Maternité Régionale
Locations (1):
- CHRU Nancy - Maternité Régionale, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided